CLINICAL TRIAL: NCT02435641
Title: A Prospective Study to Investigate Relationships Between Patient and Family Caregiver Distress Following Neuroscience ICU Admission
Brief Title: Patient and Caregiver Psychological Functioning Following Neuro-ICU Admission: A Prospective Investigation
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Clinical Psychologist, Massachusetts General Hospital
Other Study IDs: 2014P002793
Record Dates: First submitted 2015-04-29; First posted 2015-05-06 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Intensive Care Neurological Disorder
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU Questionnaires: After enrollment, all subjects (patients and their primary caregiver) will be given baseline measures assessing: sociodemographics, depression, anxiety, distress, stress, PTSD, coping, mindfulness, quality of life, satisfaction with life, resiliency/self efficacy (patient only), patient caregiver interaction, caregiver preparedness (caregiver only), caregiver self efficacy (caregiver only), quality of adherence measure, and health care satisfaction.
  Subjects will complete the same measures again at time 2 (3 months) and time 3 (6 months). The study endpoint is time 3 follow up (6 months).
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — All subjects (patients and caregivers) will complete a battery of psychological questionnaires at baseline (ICU admission), 3 months post-baseline, and 6 months post-baseline.

SUMMARY:
The current study has the following objectives:

1. To determine predictors of time 2 and 3 (3 and 6 months post-ICU admission) depression, PTSD, satisfaction with life and quality of life in both patients and caregivers, after controlling for injury severity and impairment.
2. To determine factors associated with patient and caregiver satisfaction with medical care at time 2 and time 3.

The investigators would thus be able to identify the best time point for intervention delivery, intervention targets, and risk factors for chronic psychological distress.

ELIGIBILITY:
Inclusion criteria for patients:

1. 18 years of age and older
2. English fluency and literacy
3. Admitted to the Neuro-ICU

Inclusion criteria for family caregivers:

1. 18 years of age and older
2. English fluency and literacy
3. Family member of patient who is identified by patient as the primary caregiver

Exclusion criteria:

1. Patients who cannot complete questionnaires due to their medical condition, and are anticipated to not be able to complete questionnaires at any of the future time points, due to permanent impairment.
2. Patients who lack decision-making capacity as determined by their clinical team
3. Patients who are comfort measures only (CMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Neuro-ICU and their family caregivers
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2015-03; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Change between Baseline (week 0), 3-month Follow Up (week 13) and 6-month Follow Up (week 26)
  Measures symptoms of anxiety and depression.
Posttraumatic Stress (PCL-S) | Change between Baseline (week 0), 3-month Follow Up (week 13) and 6-month Follow Up (week 26)
  Measures symptoms of posttraumatic stress disorder
Satisfaction with Life Questionnaire (SWL) | Change between Baseline (week 0), 3-month Follow Up (week 13) and 6-month Follow Up (week 26)
  Measures global cognitive judgements of satisfaction with one's life
World Health Organization QOL Questionnaire (WHOQOL-BREF) | Change between Baseline (week 0), 3-month Follow Up (week 13) and 6-month Follow Up (week 26)
  Measures one's perceptions in the context of their culture and value systems, and their personal goals, standards and concerns.

SECONDARY OUTCOMES:
General Self-Efficacy Scale | Change between Baseline (week 0), 3-month Follow Up (week 13) and 6-month Follow Up (week 26)
  Measures optimistic self-beliefs to cope with a variety of difficult demands in life. (Completed by the patient only).
Caregiver Self-Efficacy Scale | Change between Baseline (week 0), 3-month Follow Up (week 13) and 6-month Follow Up (week 26)
  Measures 3 domains of caregiving self-efficacy: Obtaining Respite, Responding to Disruptive Patient Behaviors, and Controlling Upsetting Thoughts. (Completed by the caregiver only).
Distress Thermometer Scale | Change between Baseline (week 0), 3-month Follow Up (week 13) and 6-month Follow Up (week 26)
  Measures one's distress, anxiety, depression, anger, and need for help over the past week on a scale from 0 to 10.
Visual Analog Stress Scale | Change between Baseline (week 0), 3-month Follow Up (week 13) and 6-month Follow Up (week 26)
  Measures one's distress, stress, and ability to cope with that stress over the past week on a scale from 0 to 10.
Healthcare satisfaction (CSQ-8) | Change between Baseline (week 0), 3-month Follow Up (week 13) and 6-month Follow Up (week 26)
  Measures one's satisfaction with health, human service, governmental, and public benefit programs and services.
Cognitive and Affective Mindfulness Scale (CAMS) | Change between Baseline (week 0), 3-month Follow Up (week 13) and 6-month Follow Up (week 26)
  Measures the degree to which individuals experience their thoughts and feelings.
Patient-caregiver interaction (Intimate Bond Measure) | Change between Baseline (week 0), 3-month Follow Up (week 13) and 6-month Follow Up (week 26)
  Measures the dimensions of care and control between partners in an intimate relationship.
Measure of Current Status (MOCS-A) | Change between Baseline (week 0), 3-month Follow Up (week 13) and 6-month Follow Up (week 26)
  Measures participants' current self-perceived status on several skills that are targeted by the intervention: the ability to relax at will, recognize stress-inducing situations, restructure maladaptive thoughts, be assertive about needs, and choose appropriate coping responses as needed.
Qualitative Adherence Measure | Change between Baseline (week 0), 3-month Follow Up (week 13) and 6-month Follow Up (week 26)
  Measures medication and instruction adherence amongst patients and caregivers.
Caregiving Preparedness (Preparedness for Caregiving Scale) | Change between Baseline (week 0), 3-month Follow Up (week 13) and 6-month Follow Up (week 26)
  A caregiver self-rated instrument that consists of eight items that asks caregivers how well prepared they believe they are for multiple domains of caregiving. Preparedness is defined as perceived readiness for multiple domains of the caregiving role such as providing physical care, providing emotional support, setting up in-home support services, and dealing with the stress of caregiving. (Completed by the caregiver only).

OTHER OUTCOMES:
Age, Gender, Race, Ethnicity, Marital Status, Education Status, and Employment Status of Patients/Caregivers in the ICU | Baseline (week 0)
  This questionnaire asks ICU patients/caregivers to report their age, gender, race, ethnicity, marital status, highest level of education, and primary employment status over the last 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States